CLINICAL TRIAL: NCT01766479
Title: Non-cathartic Computed Tomographic Colonography to Screen for Colorectal Neoplasia in Subjects With a Family History of Colorectal Cancer
Brief Title: Non-cathartic Computed Tomographic Colonography to Screen Subjects With a Family History of Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: MTedeschi
Record Dates: First submitted 2012-12-31; First posted 2013-01-11 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Neoplasia
Keywords: Colorectal cancer; colorectal neoplasia; CT colonography; advanced neoplasia; colonoscopy; family history
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Family Degree-relatives of pts. with CRC (Experimental): Consecutive patients admitted with CRC diagnosis (index case, IC) were prospectively evaluated. Following the systematic identification of ICs with inherited predispositions to CRC, ICs who agreed to contact their FDRs ≥40 years old were included. Available FDRs were invited to undergo non-cathartic CTC, with OC the following day.
  Interventions: Radiation: CT colonography

INTERVENTIONS:
Radiation: CT colonography

SUMMARY:
Background: Although subjects with first-degree relatives (FDR) with a history of colorectal cancer (CRC) are at increased risk for CRC, compliance to screening colonoscopy is suboptimal. Computed tomographic colonography (CTC) has been recognized as an alternative for CRC screening in average risk subjects, but less information is available on its performance in FDRs.

Aims: To prospectively assess the accuracy of CTC as a screening tool in FDRs using colonoscopy (OC) with segmental unblinding as reference standard.

Methods: Consecutive patients admitted with CRC diagnosis (index case, IC) were prospectively evaluated. Following the systematic identification of ICs with inherited predispositions to CRC, ICs who agreed to contact their FDRs ≥40 years old were included. Available FDRs were invited to undergo non-cathartic CTC, with OC the following day. Sensitivity/specificity/PPV/NPV of CTC was assessed for detecting subjects with any lesion ≥6 mm, ≥10 mm, and for advanced neoplasia ≥6 mm.

ELIGIBILITY:
Inclusion Criteria:

* Family history for CRC (first degree)
* Age >40 years old

Exclusion Criteria:

* Contraindications to colonoscopy or CT colonography
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 844 (Actual)
Dates: Start 2009-05; Primary Completion 2011-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of patients in whom colorectal polyps and colorectal neoplasia have been detected by CT colonography, by adopting colonoscopy as gold standard, as a measure of efficacy. | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico humanitas, Milan, Italy, Italy